CLINICAL TRIAL: NCT00005297
Title: Age-related Prevalence of Sleep Respiratory Disturbances
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 2020; R01HL040930 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2005-03

CONDITIONS: Lung Diseases; Heart Diseases; Hypertension; Sleep Apnea Syndromes
MeSH Terms: conditions — Lung Diseases; Heart Diseases; Hypertension; Sleep Apnea Syndromes

SUMMARY:
To determine the prevalence and longitudinal course of sleep apnea among men and women and to examine the associations of apnea, oxygen desaturation, snoring, high blood pressure, and other biomedical correlates.

DETAILED DESCRIPTION:
BACKGROUND:

Sleep apnea is characterized by repetitive cessations of respiration during sleep with consequent decreases in arterial oxygen saturation. Sleep apnea can be caused by upper airway obstruction or by central nervous system failure to sufficiently excite the diaphragm and accessory respiratory muscles. However, in most cases, both processes are involved. Hypopneas, in which airflow is significantly compromised without complete cessations of respiratory flow, and snoring are often found in association with apneas. Both apneas and hypopneas cause repetitive disruptions of sleep, consequent daytime somnolence, and complex cardio-respiratory disturbances.

DESIGN NARRATIVE:

The study was longitudinal in design. A stratified random sample of adults in San Diego was used to examine risk factors in the prevalence of sleep respiratory disturbances. A structured random sample was selected by random digit telephone dialing. Subjects were studied in their homes. Some were followed yearly during the project. Each volunteer gave a brief sleep history and medical review, including blood pressure measurement, the National Interview Survey, And Quality of Well-being Scale. Blood oxygen saturation, pulse rate, snoring, and sleep duration were recorded for three nights. State-of-the-art computerized pulse oximeters and microprocessor-based activity/light monitors were used. Subjects found to have the most severe sleep respiratory disturbances underwent laboratory polysomnograms to add descriptive data and to validate the survey methodology. The prevalence of respiratory disturbances in sleep was analyzed as a function of age and sex. Associations with several aspects of morbidity were determined. The longitudinal course of respiratory disturbances in sleep were examined.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1990-04; Study Completion 1997-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Kripke — University of California, San Diego

REFERENCES:
- [Background] Espiritu RC, Kripke DF, Ancoli-Israel S, Mowen MA, Mason WJ, Fell RL, Klauber MR, Kaplan OJ. Low illumination experienced by San Diego adults: association with atypical depressive symptoms. Biol Psychiatry. 1994 Mar 15;35(6):403-7. doi: 10.1016/0006-3223(94)90007-8. PMID 8018787
- [Background] Kripke DF, Ancoli-Israel S, Klauber MR, Wingard DL, Mason WJ, Mullaney DJ. Prevalence of sleep-disordered breathing in ages 40-64 years: a population-based survey. Sleep. 1997 Jan;20(1):65-76. doi: 10.1093/sleep/20.1.65. PMID 9130337
- [Background] Ando K, Kripke DF. Light attenuation by the human eyelid. Biol Psychiatry. 1996 Jan 1;39(1):22-5. doi: 10.1016/0006-3223(95)00109-3. PMID 8719122
- [Background] Rex KM, Kripke DF, Cole RJ, Klauber MR. Nocturnal light effects on menstrual cycle length. J Altern Complement Med. 1997 Winter;3(4):387-90. doi: 10.1089/acm.1997.3.387. PMID 9449059
- [Background] Jean-Louis G, Kripke DF, Ancoli-Israel S, Klauber MR, Sepulveda RS, Mowen MA, Assmus JD, Langer RD. Circadian sleep, illumination, and activity patterns in women: influences of aging and time reference. Physiol Behav. 2000 Jan;68(3):347-52. doi: 10.1016/s0031-9384(99)00186-9. PMID 10716544
- [Background] Jean-Louis G, von Gizycki H, Zizi F. Predictors of subjective sleepiness induced by melatonin administration. J Psychosom Res. 1999 Oct;47(4):355-8. doi: 10.1016/s0022-3999(98)00076-2. PMID 10616229
- [Background] Jean-Louis G, Mendlowicz MV, Von Gizycki H, Zizi F, Nunes J. Assessment of physical activity and sleep by actigraphy: examination of gender differences. J Womens Health Gend Based Med. 1999 Oct;8(8):1113-7. doi: 10.1089/jwh.1.1999.8.1113. PMID 10565670
- [Background] Jean-Louis G, Zizi F, von Gizycki H, Hauri P. Actigraphic assessment of sleep in insomnia: application of the Actigraph Data Analysis Software (ADAS). Physiol Behav. 1999 Jan 1-15;65(4-5):659-63. doi: 10.1016/s0031-9384(98)00213-3. PMID 10073464